CLINICAL TRIAL: NCT04182256
Title: A Prospective Study: Magnetic Spiderman for Preparation of Donor Livers' Inferior Vena Cava
Brief Title: Magnetic Spiderman for Preparation of Liver Donation
Acronym: MSPLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-2017ZD1-01
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Liver Transplant; Complications; Surgical Injury
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS group (Experimental): In the MS group, the MS grips the HVC through the magnet adsorbed onto the wall of the basin containing the liver. By changing the position of the MS on the wall of the basin, the surgeon is able to expose the surgical field.
  Interventions: Device: MS
- MA group (No Intervention): In MA group, assistants use vessel forceps to pull the HVC according to the attending's requirements.

INTERVENTIONS:
Device: MS — Magnetic Spiderman (MS) is a novel surgical instrumentIt. It consists of a circular neodymium iron boron magnet packed in a stainless-steel case with a spring and a jagged clamp, which gives it a spider-like appearance.
  Arms: MS group

SUMMARY:
Due to many vascular branches on the supra-hepatic vena cava (SHVC) and infra-hepatic vena cava (IHVC), in the whole procedures of preparation of liver donation, preparation of hepatic vena cava (HVC) is the most key and troublesome step. Magnetic Spiderman (MS) is a novel surgical instrument, designed and created to solve the vital problems of preparation of liver donation's HVC. Therefore, the aim of this study is to evaluate the feasibility and security of MS when using it prepare the liver donation's HVC.

DETAILED DESCRIPTION:
From January 1 2020 to June 30 2020, after inclusion and exclusion, donors' livers will be divided to MS group and manual (MA) group. In MS group, MS grips the SHVC and IHVC, respectively. MS's magnets are adsorbed on the wall of the basin and MS can pull the HVC accordingly. By changing the position of MS on the wall of the basin, the attending can expose the surgical field that make the operation convenient. In MA group, assistants use vessel forceps to pull the HVC according to the attending's requirements. In both groups, right adrenal vein, phrenic veins and other branches of the HVC are isolated and ligated, then SHVC and IHVC where MS's clamps gripped are cut off. After preparation, the SHVC and IHVC remain at least 1.5 cm. Excess diaphragms are removed. Outcomes of two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving donation after cardiac death in the First Affiliated Hospital, School of Medicine, Xi'an Jiaotong University.

Exclusion Criteria:

* patients whose age<18, or >60
* patients who do not have intact clinical data
* patients who are inability to participate in follow-up
* patients who undergo split liver transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The number of damaged points on HVC | measured at the time of the end of preparation HVC; up to 1 hour
  the number of damaged points on the HVC during the preparation
Operation time | measured at the time of the end of preparation HVC; up to 1 hour
  operation time of preparation of HVC
The number of assistants | measured at the time of the end of preparation HVC; up to 1 hour
  the number of assistants ensuring smooth operation according to attending's requirement
Leak test | measured at the time of the end of preparation HVC; up to 1 hour
  we use nondestructive vascular forceps to occlude the SHVC and IHVC, and perfused about 100 ml organ preservation solution through portal vein. If HVC and portal vein bulge and does not leak, the leak test is negative. Otherwise, it is positive.
HVC hemorrhage | measured at the time of liver implanted to the recipient; up to 1 hour
  Whether HVC hemorrhage after implantation

SECONDARY OUTCOMES:
Frequency of MS's detachment | measured at the time of the end of preparation HVC; up to 1 hour
  the frequency of MS's detachment from the vasculature and basin wall.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No